CLINICAL TRIAL: NCT03786081
Title: A Phase 1b/2 Open-Label Trial of Tisotumab Vedotin (HuMax®-TF-ADC) Monotherapy and in Combination With Other Agents in Subjects With Recurrent or Stage IVB Cervical Cancer
Brief Title: Safety and Efficacy of Tisotumab Vedotin Monotherapy & in Combination With Other Cancer Agents in Subjects With Cervical Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Genmab (Industry); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Belgian Gynaecological Oncology Group (Other); GOG Foundation (Network); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCT1015-05; InnovaTV 205 (Other: Genmab); MK-3475-834 (Other: Merck Sharp & Dohme LLC); ENGOT-cx8 (Other: European Network of Gynaecological Oncological Trial); GOG-3024 (Other: GOG Foundation); KEYNOTE-834 (Other: Merck Sharp & Dohme LLC); 2017-004758-40 (EudraCT Number)
Record Dates: First submitted 2018-12-13; First posted 2018-12-24 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer
Keywords: cervical carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — tisotumab vedotin; Bevacizumab; pembrolizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- A: Tisotumab Vedotin + bevacizumab (Experimental): Dose escalation: Tisotumab vedotin in combination with bevacizumab once every three weeks in previously treated patients
  Interventions: Drug: Tisotumab Vedotin; Drug: Bevacizumab
- B: Tisotumab vedotin + pembrolizumab (Experimental): Dose escalation: Tisotumab vedotin in combination with pembrolizumab once every three weeks in previously treated patients
  Interventions: Drug: Tisotumab Vedotin; Drug: Pembrolizumab
- C: Tisotumab vedotin + carboplatin (Experimental): Dose escalation: Tisotumab vedotin in combination with carboplatin once every three weeks in previously treated patients
  Interventions: Drug: Tisotumab Vedotin; Drug: Carboplatin
- D: Tisotumab vedotin + carboplatin (Experimental): Dose expansion:Tisotumab vedotin in combination with carboplatin once every three weeks in previously untreated patients
  Interventions: Drug: Tisotumab Vedotin; Drug: Carboplatin
- E: Tisotumab vedotin + pembrolizumab (Experimental): Dose expansion: Tisotumab vedotin in combination with pembrolizumab once every three weeks in previously untreated patients
  Interventions: Drug: Tisotumab Vedotin; Drug: Pembrolizumab
- F: Tisotumab vedotin + pembrolizumab (Experimental): Dose expansion: Tisotumab vedotin in combination with pembrolizumab once every three weeks in previously treated patients
  Interventions: Drug: Tisotumab Vedotin; Drug: Pembrolizumab
- G: Tisotumab vedotin monotherapy (Experimental): Dose expansion: Tisotumab vedotin monotherapy weekly for three weeks and 1 week off (28 day treatment cycle) in previously treated patients.
  Interventions: Drug: Tisotumab Vedotin
- H: Tisotumab vedotin + pembrolizumab + carboplatin +/- bevacizumab (Experimental): Dose expansion: Tisotumab vedotin in combination with pembrolizumab and carboplatin with or without bevacizumab once every three weeks in previously untreated patients
  Interventions: Drug: Tisotumab Vedotin; Drug: Bevacizumab; Drug: Pembrolizumab; Drug: Carboplatin

INTERVENTIONS:
Drug: Tisotumab Vedotin — Given into the vein (IV)
  Other Names: TIVDAK
Drug: Bevacizumab — Given via IV
  Other Names: Avastin
  Arms: A: Tisotumab Vedotin + bevacizumab; H: Tisotumab vedotin + pembrolizumab + carboplatin +/- bevacizumab
Drug: Pembrolizumab — Given via IV
  Other Names: KEYTRUDA®
  Arms: B: Tisotumab vedotin + pembrolizumab; E: Tisotumab vedotin + pembrolizumab; F: Tisotumab vedotin + pembrolizumab; H: Tisotumab vedotin + pembrolizumab + carboplatin +/- bevacizumab
Drug: Carboplatin — Given via IV
  Other Names: Paraplatin
  Arms: C: Tisotumab vedotin + carboplatin; D: Tisotumab vedotin + carboplatin; H: Tisotumab vedotin + pembrolizumab + carboplatin +/- bevacizumab

SUMMARY:
This is an open label, multi-center trial of tisotumab vedotin monotherapy and in combination with bevacizumab, pembrolizumab, or carboplatin in subjects with recurrent or stage IVB cervical cancer.

The trial consists of two-parts a dose escalation part and an expansion part. The expansion part of the trial will be initiated once the Recommended Phase 2 Dose (RP2D) of the combinations have been determined in the dose escalation part.

DETAILED DESCRIPTION:
The dose escalation part will occur in participants with cervical cancer who have progressed during or after standard of care therapy and who are intolerant or ineligible to receive standard of care treatments. Arm A will be conducted by escalating doses of both tisotumab vedotin and bevacizumab. Dose escalations of the tisotumab vedotin + pembrolizumab and tisotumab vedotin + carboplatin combinations (Arms B and C, respectively) will be conducted by combining fixed doses of either pembrolizumab or carboplatin with increasing doses of tisotumab vedotin.

The dose expansion part of this study (Arms D through H) will be conducted in 2 populations: participants with cervical cancer who have not received prior systemic therapy for recurrent or stage IVB cervical cancer (Arms D, E, and H) and participants with cervical cancer who have progressed on or after at least 1 but no more than 2 prior systemic therapies (Arms F and G).

Participants enrolled to Arms D, E, F and H will receive the RP2D of tisotumab vedotin established in the dose escalation part. Participants enrolled to Arm G will receive tisotumab vedotin weekly (at a dose lower than subjects in all other Arms) for three weeks and 1 week off (28-day treatment cycle).

ELIGIBILITY:
Inclusion Criteria:

* Must have squamous, adenosquamous, or adenocarcinoma of the cervix and progressed on or after standard of care treatments or are ineligible or intolerant to standard of care for recurrent or stage IVB cervical cancer (Arms A, B and C only).
* Must have squamous, adenosquamous, or adenocarcinoma of the cervix and must not have received prior systemic therapy for recurrent or stage IVB cervical cancer (Arms D, E, and H only).
* Must have squamous, adenosquamous, or adenocarcinoma of the cervix and progressed on or after at least one but no more than two prior systemic therapies for recurrent or stage IVB cervical cancer (Arms F and G only).
* Must have baseline measurable disease per RECIST v1.1.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (All Arms).
* Is not pregnant, breastfeeding, or expecting to conceive children within the projected duration of the trial and for at least 6 months after the last trial treatment administration
* Participants of childbearing potential must agree to use adequate contraception during and for 6 months after the last dose of trial treatment administration.
* Must sign an informed consent form (ICF) indicating the trial subject understands the purpose of and procedures required for the trial and are willing to participate in the trial (All Arms).

Exclusion Criteria:

* Has clinically relevant bilateral hydronephrosis which cannot be alleviated by ureteral stents or percutaneous drainage. (All Arms)
* Has clinical signs or symptoms of gastrointestinal obstruction and requires parenteral hydration and/or nutrition. Post-operative obstructions within 4 weeks of abdominal surgery are permitted. (All Arms)
* Has clinically significant bleeding issues or risks

  * Prior history (within 3 months) or current evidence of hemoptysis (1/2 teaspoon or more) (Arm A and bevacizumab-eligible participants in Arm H)
  * Recent (within 4 weeks of first dose of trial treatment) clinically significant gastrointestinal or vaginal bleeding requiring PRBC transfusion (Arms A and H only)
  * Recent (within 4 weeks of first dose of trial treatment) evidence of wound healing complications that require medical intervention (Arms A and H only)
* Has active ocular surface disease at baseline. Subjects with prior history of cicatricial conjunctivitis are ineligible (All Arms).
* Clinically significant cardiac disease
* Requires anti-coagulation therapy (Arms A and H only)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Dose escalation: Dose Limiting Toxicities (DLTs) | DLTs will be identified during the first treatment cycle (21 day cycles)
  To establish the MTD and RP2D of tisotumab vedotin in combination
Dose expansion: Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | approximately 2 years
  Objective response is defined as confirmed partial response (PR) or complete response (CR)

SECONDARY OUTCOMES:
Number of adverse events (AEs) | up to 2 years
  Any untoward medical occurrence in a clinical trial participant whether or not considered related to the medicinal product.
Dose escalation: ORR per RECIST v1.1 | approximately 2 years
  Objective response is defined as confirmed PR or CR.
Duration of Response (DOR) per RECIST v1.1 by investigator assessment | approximately 2 years
  Will be calculated from the date of initial documentation of a response (CR or PR) to the date of first documented evidence of progressive disease (PD) or death.
Time to Response (TTR) per RECIST v1.1 by investigator assessment | approximately 2 years
  Will be calculated from the date of the first dose to the date of the initial documentation of response (CR or PR).
Progression free survival (PFS) per RECIST v1.1 by investigator assessment | approximately 2 years
  The time from the date of the first trial drug administration to the date of the first documented disease progression or death due to any cause.
Overall Survival (OS) | approximately 2 years
  The time from the date of the first trial drug administration to the date of death due to any cause.
Maximum concentration (Cmax) (All Arms except G) | Up to 42 days
  Pharmacokinetic (PK) parameter
Cmax (Arm G only) | Up to 2 years
  PK parameter
Trough Concentration (Ctrough) (All Arms) | Up to 2 years
  PK parameter
Area under the concentration-time curve (AUC) (All Arms except G) | Through 21 days after first dose
  PK parameter
AUC (Arm G only) | Through 8 days after first dose
  PK parameter
Anti-drug antibodies (ADAs) | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (68):
- United States (24):
  - Arizona Oncology Associates, Phoenix, Arizona
  - Univ California, Irvine Medical Center, Orange, California
  - Olive View - UCLA Research and Education Institute, Sylmar, California
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Augusta University, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center, Westwood, Kansas
  - Oschner Clinic, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Billings Clinic Cancer Center, Billings, Montana
  - Montana Cancer Consortium, Billings, Montana
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - University of Cincinnati Physicians Group, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Hilliard, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Brown University - Women's and Infant Hospital, Providence, Rhode Island
  - St Francis Hospital Cancer Center, Greenville, South Carolina
  - Huntsman Cancer Center, Salt Lake City, Utah
  - Carilion Clinic, Roanoke, Virginia
- Belgium (12):
  - AZ Sint-Jan, Bruges
  - Cliniques universitaires Saint-Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Universitair Ziekenhuis Antwerpen (UZA), Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - Universitaire Ziekenhuizen Leuven,, Leuven
  - Centre Hospitalier de l'Ardenne, Libramont
  - Centre Hospitalier Universitaire (CHU) de Liège, Liège
  - Grand Hôpital de Charleroi, Loverval
  - CHU UCL Namur, Namur
  - Sainte-Elisabeth, Namur
- Czechia (5):
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice Bulovka, Prague
  - Nemocnice Na Bulovce, Prague
- Rigshospitalet, Copenhagen, Denmark
- Ireland (4):
  - Cork University Hospital, Cork
  - Mater Misericordiae University Hospital, Dublin
  - Waterford Regional Hospital, Waterford
  - University Hospital Waterford, Waterford
- Italy (5):
  - Azienda Ospedaliera Cannizzaro, Catania
  - IEO Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Netherlands (8):
  - Amsterdam UMC, Locatie AMC, Amsterdam
  - AMC Medical Research, Amsterdam
  - Universitair Medisch Centrum Groningen (UMCG), Groningen
  - Radboudumc, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Erasmus University Medical Center Rotterdam, Rotterdam
  - UMC Utrecht, Utrecht
  - University Medical Center Utrecht (UMC Utrecht), Utrecht
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital 12 De Octubre, Madrid
- Turkey (Türkiye) (2):
  - Baskent University Adana Application and Research Center, Adana
  - Baskent University Ankara Hospital, Ankara
- United Kingdom (3):
  - Velindre Cancer Centre, Cardiff, South Glamorgan
  - Beatson West of Scotland Cancer Centre, Glasgow, Strathclyde
  - Royal Marsden Hospital- Sutton, Sutton, Surrey

REFERENCES:
- [Derived] Vergote I, Van Nieuwenhuysen E, O'Cearbhaill RE, Westermann A, Lorusso D, Ghamande S, Collins DC, Banerjee S, Mathews CA, Gennigens C, Cibula D, Tewari KS, Madsen K, Kose F, Jackson AL, Boere IA, Scambia G, Randall LM, Sadozye A, Baurain JF, Gort E, Zikan M, Denys HG, Ottevanger N, Forget F, Mondrup Andreassen C, Eaton L, Chisamore MJ, Viana Nicacio L, Soumaoro I, Monk BJ. Tisotumab Vedotin in Combination With Carboplatin, Pembrolizumab, or Bevacizumab in Recurrent or Metastatic Cervical Cancer: Results From the innovaTV 205/GOG-3024/ENGOT-cx8 Study. J Clin Oncol. 2023 Dec 20;41(36):5536-5549. doi: 10.1200/JCO.23.00720. Epub 2023 Aug 31. PMID 37651655